CLINICAL TRIAL: NCT01592942
Title: A Randomized Multi-center Study of Tissue Glue Fixation of Optilene™ Mesh With Histoacryl™ or Self-gripping Parietex ProGrip™ Compared to Conventional Non-absorbable Suture Fixation of Ultrapro™ Mesh
Brief Title: Mesh Fixation in Lichtenstein Hernioplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kuopio University Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other); Paijat-Hame Hospital District (Other); North Karelia Central Hospital (Other); East Savo Hospital District (Other)
Responsible Party: Principal Investigator, Hannu Paajanen, PhD, MD, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KUH5200627; KUH 31//2012 (Registry Identifier: KUH 31//2012)
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Inguinal Hernia
Keywords: inguinal hernia; mesh fixation; glue; Lichtenstein
MeSH Terms: conditions — Hernia, Inguinal | interventions — Sutures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- glue fixation (Experimental): Optilene™ mesh 60 g/m2 (B. Braun), fixation Histoacryl™ cyanoacrylate glue (price 14+37 euros)
  Interventions: Device: Histoacryl
- self-gripping (Active Comparator): ProGrip™ mesh 60 g/m2 (Covidien, USA) (price 113 euros)
  Interventions: Device: Progrip
- suture fixation (Active Comparator): Ultrapro™ mesh 28 g/m2 (Ethicon, USA) (price 45 euros) fixated by non-absorbable sutures
  Interventions: Device: sutures (prolene 3-0)

INTERVENTIONS:
Device: Histoacryl — cyanoacrylate glue fixation of mesh 1 ml
  Other Names: Histoacryl glue
  Arms: glue fixation
Device: Progrip — self-gripping mesh
  Other Names: Parietex Progrip
  Arms: self-gripping
Device: sutures (prolene 3-0) — non-absorbable suture fixation 3-0
  Other Names: prolene 3-0
  Arms: suture fixation

SUMMARY:
This is a prospective, randomized multi-centre study to find out most safe, feasible, painless and cost-effective mesh fixation method in inguinal hernia operation. Three mesh fixation techniques are compared to find out best technique in local anaesthesia Lichtenstein operation. Our hypothesis is that glue fixation is safe, simple and cheap method compared to conventional Lichtenstein technique.

DETAILED DESCRIPTION:
Some 650 patients with inguinal hernia are operated using Lichtenstein operation in local anaesthesia. Mesh fixation is performed using 3 methods: Optilene™ mesh + cyanoacrylate glue (n=200), self-fixing Parietex Progrip™ mesh (n=200) and non-absorbable sutures with Ultrapro™ mesh (n=200). Operative time and pain scores, immediate postoperative outcome, quality-of-life and total costs are followed 1, 7, 30 days and 1 and 5 years postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* primary or recurrent inguinal hernia
* unilateral or bilateral

Exclusion Criteria:

* femoral hernia
* massive scrotal hernia
* allergy to polypropylene
* patient's refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2012-08; Primary Completion 2019-03 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
pain | 5 years
  pain scores (VAS 0-10) preoperatively and after surgery

SECONDARY OUTCOMES:
costs | 1 year
  operative cost-effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Hannu EK Paajanen, MD, PhD, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Finland